CLINICAL TRIAL: NCT00660959
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Lixivaptan Capsules in Subject With Euvolemic Hyponatremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry); Biogen (Industry)
Responsible Party: Cardiokine, Inc, Cardiokine, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CK-LX3405
Record Dates: First submitted 2008-04-15; First posted 2008-04-18 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-11

CONDITIONS: Hyponatremia With Normal Extracellular Fluid Volume
Keywords: Euvolemic; Hyponatremia; Serum Sodium; Fluid Overload; Vasopressin Antagonist
MeSH Terms: conditions — Hyponatremia; Edema | interventions — lixivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator (Experimental): lixivaptan
  Interventions: Drug: lixivaptan
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lixivaptan — oral capsule
  Arms: Active Comparator
Drug: placebo — oral capsule
  Arms: Placebo

SUMMARY:
The present study is designed to confirm and extend the observation from previous studies that lixivaptan therapy corrects hyponatremia, in euvolemic subject, including subjects with SIADH.

DETAILED DESCRIPTION:
Phase I Phase II clinical trials have demonstrated that lixivaptan may play an important role in treating hyponatremia and the signs and symptoms of water retention associated with HF, liver cirrhosis with ascites (LCWA) and syndrome of inappropriate antidiuretic hormone (SIADH). Lixivaptan was previously evaluated in disease states characterized by hyponatremia with euvolemia (SIADH)and hyponatremia combined with fluid overload (HF, LCWA). Lixivaptan resulted in correction in hyponatremia together with a marked aquaresis in subject with volume overload. The present study is designed to confirm and extend the observation from previous studies that lixivaptan therapy corrects hyponatremia, in euvolemic subject, including subjects with SIDH.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men or women aged 18 or older
* Diagnosis of euvolemic hyponatremia (120 ≤ Na+<130 mEq/L)
* Hospitalized or willing to be admitted to a monitored setting for approximately the first 48 hours of treatment

Exclusion Criteria:

* Pregnant or breast-feeding women, or women planning to become pregnant or to breastfeed
* Symptomatic hyponatremia (e.g., lethargy, coma, seizures, changes in mental status attributable to hyponatremia)
* Acute or transient hyponatremia (e.g., associated with head trauma or postoperative state)
* Hyponatremia in hypovolemic states. Hypovolemic hyponatremia is defined as the presence of clinical evidence of extracellular fluid volume depletion
* Hyponatremia as a result of any medication that can safely be withdrawn
* Hyponatremia due to hypothyroidism or adrenal insufficiency
* Diagnosis of psychogenic polydipsia
* Receiving within 7 days of enrollment, other medication for treatment of hyponatremia specifically: demeclocycline, lithium carbonate, urea, or conivaptan
* Use of radiotherapy and chemotherapy within 2 wks of randomization
* Likely to require, or to receive IV saline for correction of symptomatic or asymptomatic severe hyponatremia during the course of the study
* Supine systolic arterial blood pressure of ≤ 90 mmHg
* Serum creatinine >3.0 mg/dL
* History of uncontrolled type 2 diabetes mellitus
* Severe pulmonary artery hypertension: patients whose condition is expected to deteriorate with sudden shifts in fluid volumes and cardiac filling pressures
* Established diagnosis of New York Heart Association (NYHA) class III or IV heart failure
* History of myocardial infarction, unstable angina or evidence of active ischemia within 30 days prior to screening
* History of cerebral vascular accident (CVA) within 60 days prior to screening
* Established diagnosis of nephrotic syndrome
* Advanced liver disease or documented diagnosis of cirrhosis or alcoholic hepatitis
* Urinary tract obstruction (benign prostatic hypertrophy [BPH] allowed if non-obstructive)
* History of alcohol abuse or illicit drug use within the past 6 months
* Terminally ill or moribund condition with little chance of short-term survival
* Receiving vasopressin or its analogs for treatment of any condition
* Known allergy to any vasopressin antagonist
* Previous participation in a lixivaptan study
* Recipient of any investigational treatment (drug or device) within 30 days prior to baseline visit
* Unable to take oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Average daily area under the curve (AUC) of change from baseline in serum sodium concentrations up to 72 hrs in lixivaptan treated subjects compared to placebo | 60 days

SECONDARY OUTCOMES:
Change from baseline in serum sodium on Day 30 | 60 days
Percentage of subjects achieving normalized serum sodium (Na+ ≥ 135 mEq/L) | 60 days
Time to first normalization of serum sodium (Na+≥135 mEq/L) | 60 days

CONTACTS AND LOCATIONS:
Locations (68):
- United States (37):
  - Research Site 1, Mobile, Alabama
  - PsyPharma Global, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site 1, Los Angeles, California
  - Research Site 1, Roseville, California
  - Research Site, Aurora, Colorado
  - The George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Healthcare Clinical Data, Inc, North Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Research Site, Augusta, Georgia
  - RTR Medical Group, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site 1, Iowa City, Iowa
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Research Site, Belmont, Massachusetts
  - Research Site, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Research Site, Kansas City, Missouri
  - Research Site 1, Las Vegas, Nevada
  - Research Site 1, Albany, New York
  - Erie County Medical Center, Buffalo, New York
  - Research Site, New York, New York
  - Three Rivers Health and Rehabilitation, Windsor, North Carolina
  - Atrium Medical Center, Middletown, Ohio
  - Kettlie Joseph Daniels MD, Inc, Toledo, Ohio
  - Research Site 1, Camp Hill, Pennsylvania
  - Research Site 1, Doylestown, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site 1, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site 1, Columbia, South Carolina
  - SunStar Geriatrics Healthcare, Georgetown, Texas
  - Clinical Trial Network, Houston, Texas
  - Aspen Clinical Research, Orem, Utah
  - The Glennan Center for Geriatrics and Gerontology, Norfolk, Virginia
  - Internal Medicine Northwest, Tacoma, Washington
- Belgium (2):
  - UZ Gasthulsberg, Leuven
  - Centre Hospitalier de Tubize, Tubize
- Canada (3):
  - Research SIte, Greenfield Park, Quebec
  - Research Site 1, Montreal, Quebec
  - Research Site, Montreal, Quebec
- Germany (9):
  - Research Site, Dresden, Germany
  - Research Site, Hanover, Hannover
  - Research Site, Magdeburg, Magdeburg
  - Research Site, Berlin
  - Research Site, Giessen
  - Research Site, Heidelberg
  - Research SIte, Konstanz
  - Research Site, München
  - Research Site, Würzburg
- India (6):
  - Baby Memorial Hospital, Calicut, Kerala
  - Poona Hospital and Research Centre, Pune, Maharashtra
  - Vidya Sagar Institute of Mental Health and Neurosciences, New Delhi, New Delhi
  - Sir Ganga Ram Hospital, Old Rajinder Nagar, New Delhi
  - Deenanath Mengeshkar Hospital & Research Centre, Erandawane, Pune
  - Fortis Escorts Hospital, Jaipur, Rajasthan
- Poland (11):
  - Research Site 1, Podlaski, Poland
  - Research Site 1, Warsaw, Poland
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość, Zamosc
  - Research Site, Bydgoszcz
  - Research Site 1, Ciechanów
  - Research Site, Katowice
  - Research Site 1, Lodz
  - Research Site, Lublin
  - Research Site 1, Warsaw
  - Research Site, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotney, Wilgury, Łódź Voivodeship